CLINICAL TRIAL: NCT01337752
Title: A Double-blind, Placebo-controlled, Randomized Phase 2 Study of BHQ880, an Anti-Dickkopf1 (DKK1) Monoclonal Antibody (mAb), in Patients With Untreated Multiple Myeloma and Renal Insufficiency
Brief Title: Study in Patients With Untreated Multiple Myeloma and Renal Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBHQ880A2203; 2009-010875-26 (EudraCT Number)
Record Dates: First submitted 2011-04-12; First posted 2011-04-19 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma; Renal Insufficiency
Keywords: multiple myeloma; renal insufficiency; untreated multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — BHQ880; Bortezomib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- BHQ880 + bortezomib and dexamethasone (Experimental)
  Interventions: Drug: BHQ880; Drug: bortezomib; Drug: dexamethasone
- BHQ880 Placebo + bortezomib and dexamethasone (Placebo Comparator)
  Interventions: Drug: BHQ880 Placebo; Drug: bortezomib; Drug: dexamethasone

INTERVENTIONS:
Drug: BHQ880
  Arms: BHQ880 + bortezomib and dexamethasone
Drug: BHQ880 Placebo — Intravenous infusion
  Arms: BHQ880 Placebo + bortezomib and dexamethasone
Drug: bortezomib — intravenous injection
Drug: dexamethasone — Oral

SUMMARY:
The study will evaluate the effects of BHQ880 in patients with previously untreated multiple myeloma and renal insufficiency who are not considered candidates for bisphosphonate therapy. The primary objective of the study will be to evaluate the effect of BHQ880 in combination with bortezomib and dexamethasone, compared to placebo administered with the combination on the time to first Skeletal Related Event (SRE) on study.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of multiple myeloma
2. Life expectancy of more than 6 months in the absence of intervention
3. Must not have received previous or be receiving current antimyeloma therapies
4. Renal insufficiency
5. Recovered from the effects of any prior surgery or radiotherapy

Exclusion Criteria:

1. Prior IV bisphosphonate therapy at any time or oral bisphosphonate therapy within 4 months of study entry
2. Paget's disease of bone or uncorrected hyperparathyroidism
3. Impaired cardiac function
4. Known HIV, known active hepatitis B, or known or suspected hepatitis C infection
5. Pregnant or nursing (lactating) women,
6. Women of child-bearing potential, UNLESS agreeable to using 2 birth control methods

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
effect of BHQ880 compared with placebo on time to first Skeletal Related Event (SRE) in patients with untreated multiple myeloma and renal insufficiency in combination with bortezomib and dexamethasone | 18-month median time to first SRE assumed for the placebo arm
  Time to first SRE from randomization

SECONDARY OUTCOMES:
safety and tolerability of BHQ880 in combination with bortezomib and dexamethasone | From screening through month 17
  Number of patients with adverse events/serious adverse events, abnormal clinical laboratory values, and the assessment of immunogenicity
Characterize the PharmacoKinetics (PK) profiles of BHQ880 and bortezomib | At screening and weeks 1, 2, 4, 7, 10, 11, 13, 16, 25 and 34
  Determine the pharmacokinetic parameters for BHQ880 and bortezomib (Cmax, Tmax, AUC0-tlast, t1/2, and accumulation ratio of BHQ880).
Evaluate the effect of BHQ880 on bone metabolism | At screening and at months 3, 6, 12, and 18
  1) Change in bone mineral density, measured by dual-emission X-ray absorptiometry (DXA), from randomization to 12 and 18 months; 2) Change in bone strength, measured by quantitative computed tomography (qCT), from randomization to 3 and 6 months
Determine the antimyeloma effect of BHQ880 compared to placebo when used in combination with bortezomib and dexamethasone. | From the first dose of study medication through month 17
  1) The overall response rate (partial response plus complete response); 2) Progression-free survival following initiation of BHQ880

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (2):
  - University Chicago Hospital Dept. of Univ of Chicago (2), Chicago, Illinois
  - Medical Oncology Associates, PS, Spokane, Washington
- Spain (2):
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- United Kingdom (4):
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Southampton

REFERENCES:
- See also: Results for CBHQ880A2203 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=11143